CLINICAL TRIAL: NCT05950503
Title: Single-center Ambispective Observational Study on the Role of Magnetic Resonance Imaging (MRI) in the Evaluation of Patient Affected by Hepatic Metastases of Carcinoma of the
Brief Title: Role of MRI in the Evaluation of Hepatic Metastases of Colorectal Cancer
Acronym: RMN-CRC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5829
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mCRC patients: Patients with mCRC with liver-only metastases
  Interventions: Radiation: Hepatic MRI

INTERVENTIONS:
Radiation: Hepatic MRI — The patients will undergo hepatic MRI in pre-established timepoints

SUMMARY:
This study wants to evaluate the use of MRI in the managemente of mCRC with liver only metastases.

DETAILED DESCRIPTION:
This study wants to evaluate the use of MRI in the managemente of mCRC with liver only metastases.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Histological diagnosis of colorectal cancer;
* Presence of liver metastases in the staging exams (chest-abdomen CT with contrast medium or PET-CT with 18-FDG);
* At least one measurable liver lesion according to RECIST 1.1 criteria;
* Adequate organ and marrow function.

Exclusion Criteria:

* Age < 18 years;
* Inability to undergo MRI;
* Major contraindications to liver surgery;
* No written informed consent.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients with liver metastases treated at the U.O.C. of Medical Oncology of Foundation Agostino Gemelli University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
Surgery conversion rates | 3 years
  Negative conversion rate is: patients initially considered operable and subsequently not considered suitable for surgery compared to the total number of patients enrolled.
  Positive conversion rate is: patients initially deemed ineligible for surgery and subsequently operated, compared to the total number of patients enrolled.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Time from enrollment to death

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Salvatore, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Policlinico Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No